CLINICAL TRIAL: NCT06440980
Title: A Multiple-Dose Study to Investigate the Bioequivalence of Orforglipron (LY3502970) Capsules and Orforglipron Tablets in Participants With Obesity or Overweight Who Are Otherwise Healthy.
Brief Title: A Study to Compare Tablets and Capsules of Orforglipron (LY3502970) in Healthy Participants Who Are Obese or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18617; J2A-MC-GZPI (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy; Obese; Overweight; Obesity
Keywords: Pharmacokinetics
MeSH Terms: conditions — Obesity; Overweight | interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Relative bioavailability study: Cohort 1 and 2: Orforglipron (Experimental): Participants will receive different sequences of orforglipron doses administered as either tablet or capsule at different dose levels.
  Interventions: Drug: Orforglipron
- Part B: BE (bioequivalence) study: Cohort 1 and 2: Orforglipron (Experimental): Participants will receive different sequences of orforglipron doses administered as either tablet (different dose levels) or capsule (test dose levels 1 to 6).
  Interventions: Drug: Orforglipron

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970

SUMMARY:
The main purpose of this study is to see how much of orforglipron (study drug) gets into the bloodstream and how long it takes the body to get rid of it when given as capsules compared to tablets in healthy overweight and obese participants. The safety and tolerability (side effects) of orforglipron when given as capsules and tablets will also be evaluated.

The study will be conducted in two parts, with part A and B lasting up to approximately 25 and 22 weeks each respectively, including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical history and physical examination.
* Have a stable body weight for one month prior to screening (less than or equal to 5 percent body weight gain or loss) and Body Mass Index (BMI) in range of 27 to 40 kilogram per meter square (kg/m²).
* Participants must be reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have venous access sufficient to allow for blood sampling.

Exclusion Criteria:

* Have hemoglobin A1c (HbA1c) level of 6.5 percent (%) or greater.
* Have a history of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders or other significant active, uncontrolled medical conditions.
* Have significant history of or currently have major depressive disorder or psychiatric disorder within the last 2 years.
* Obesity induced by other endocrine disorders, such as Cushing's syndrome or Prader-Willi syndrome.
* Have known clinically significant gastric emptying abnormality.
* Have undergone bariatric surgery (for example: Lap-Band, Gastric Bypass)
* Have a known self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or any form of thyroid cancer.
* Have an abnormal 12-lead electrocardiogram (ECG) at screening.
* Have history of pancreatitis.
* Judged by the study investigator to be at serious suicidal risk and have answered "Yes" to either question 4 or 5 on the Columbia-Suicide Severity Rating Scale [C-SSRS]).
* Have difficulty swallowing capsules or tablets.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Part B: Pharmacokinetics (PK): Steady-state area under the concentration versus time curve from time 0 to τ hour time point AUC(0-τ) of Orforglipron capsule at test dose levels 2,3,4 and 6 along with the corresponding tablet dose strengths | Day 1 up to Week 9 (Cohort 1), Week 15 (Cohort 2)
  τ is 24 hours for once daily (QD) dosing
Part B: PK: Steady-state Maximum Observed Concentration (Cmax) of Orforglipron capsule at test dose levels 2,3,4 and 6 along with the corresponding tablet dose strengths | Day 1 up to Week 9 (Cohort 1), Week 15 (Cohort 2)

SECONDARY OUTCOMES:
Part B: PK: Steady-state AUC(0-τ) of Orforglipron capsule at test dose levels 1 and 5 along with the corresponding tablet dose strengths | Day 1 up to Week 9 (Cohort 1), Week 15 (Cohort 2)
  τ is 24 hours for QD dosing
Part B: PK: Steady-state Cmax of Orforglipron capsule at test dose levels 1 and 5 along with the corresponding tablet dose strengths | Day 1 up to Week 9 (Cohort 1), Week 15 (Cohort 2)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Altasciences Company Inc., Overland Park, Kansas
  - QPS, Springfield, Missouri
  - Fortrea Clinical Research Unit, Dallas, Texas
  - Fortrea Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Compare Tablets and Capsules of Orforglipron (LY3502970) in Healthy Participants Who Are Obese or Overweight — https://trials.lilly.com/en-US/trial/495475